CLINICAL TRIAL: NCT01956695
Title: Phase II Study Evaluating the Efficacy of Lenalidomide in Association With Rituximab in Refractory or Relapse of Primary Central Nervous System Lymphoma (PCNSL)
Brief Title: Efficacy of Lenalidomide With Rituximab in Refractory or Relapse of Primary Central Nervous System Lymphoma
Acronym: REVRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Centre Hospitalier Universitaire, Amiens (Other); Institut Bergonié (Other); University Hospital, Clermont-Ferrand (Other); University Hospital, Lille (Other); Central Hospital, Nancy, France (Other); Groupe Hospitalier Pitie-Salpetriere (Other); Centre Henri Becquerel (Other); University Hospital, Tours (Other); Centre Leon Berard (Other); University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2012-05; 2012-003786-17 (EudraCT Number)
Record Dates: First submitted 2013-09-24; First posted 2013-10-08 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2019-07

CONDITIONS: Lymphoma; Relapse
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide & Rituximab (Experimental): Induction treatment : Lenalidomide 20 mg capsule on days 1 to 21 days of a 28 days cycle for the first cycle followed by 25 mg on daily on days 1 to 21 of a 28 days cycle for cycles 2 to 8 (in the absence of hematologic toxicity. Rituximab at day 1 of each induction course 375 mg/m² intravenous.
  Maintenance : Lenalidomide 10 mg capsule on days 1 to 21 days of a 28 days cycle for 1 year or until progression or intolerance.
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid®
Drug: Rituximab
  Other Names: Mabthera®

SUMMARY:
Because Primary Central Nervous System Lymphoma (PCNSL) are mainly diffuse large B-cell lymphoma of the activated B cells (ABC) type, the investigators hypothesize that the synergy of lenalidomide with rituximab shown in systemic non-Hodgkin's lymphoma (NHL) could be observed in PCNSL.

This study will assess the efficiency of the the combination of lenalidomide and rituximab in relapsed/refractory PCNSL, and the efficiency of a maintenance treatment with lenalidomide alone in maintaining the response.

DETAILED DESCRIPTION:
The investigators use a two-stage Fleming's design based on the following hypotheses under treatment: 10% (null hypothesis, minimal clinical benefit rate), 30% (alternative hypothesis, acceptable clinical benefit rate), 3% type I error rate, 5% type II error rate. Under these hypotheses, a total of 45 assessable patients will be necessary: 22 for the first stage + 23 for the second stage.

Stage 1: following the inclusion of the first 22 assessable patients, if 0 or 1 patient has an objective response (CR, Complete Response + uCR, unconfirmed Complete Response + PR, Partial Response) at the end of induction treatment, the study would be terminated early and the treatment will be considered ineffective. If 2 or more patients have an objective response at the end of induction treatment, then the treatment will be considered as effective in this indication. Otherwise, the second group of 23 patients will be recruited.

Stage 2: if at the end of recruitment, 8 or less patients have an objective response, the investigators will conclude to inefficacy, and if 9 or more patients have an objective response, then the treatment will be considered as effective and need further exploration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old with a refractory or relapse PCNSL and who have previously received at least high dose methotrexate (> 1.5 g/m²) and high dose cytarabine (2 g/m²).
2. Patients can have received radiotherapy or intensive chemotherapy with hematopoietic stem cell rescue as part of treatment of the PCNSL or IOL
3. Patients over 18 years old with a refractory or relapse IOL and who have received either intravenous high dose methotrexate (> 1.5 g/m2) or intraocular methotrexate
4. Life expectancy > 2 months
5. Able to swallow capsules (stomach tube not allowed)
6. Adequate bone marrow function with absolute leukocytes > 2000/mm3, neutrophil count (ANC) > 1000/mm3, haemoglobin > 8 g/dl and platelets > 100 000/mm3
7. Adequate liver function with Serum SGOT/AST or SGPT/ALT < 3.0 X Upper Limit of Normal ULN ; bilirubin < 1.5 X LNS (excepted in case of hemolytic anemia or Gilbert's syndrome)
8. Calculated creatinine clearance > 40 ml/min. Patients with calculated creatinine clearance between 40 and 50ml/min lenalidomide dose will be adjusted as follows (10mg once daily)
9. Patient aged 18 years old or more and without measure of legal protection
10. Able to understand teratogenic risks of the treatment
11. Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study for at least four weeks before starting study drug, while participating in the studyand for at least 4 weeks after discontinuation of Lenalidomide and 1 year after Rituximab.. Pregnancy tests (serum β-HCG dosage) will be negative at baseline and during the study. Men must agree not to procreate a child and use condoms if their partner can procreate, during all the treatment period, during dose interruptions and for at least 4 weeks after study drug discontinuation.
12. Signed inform consent

Exclusion Criteria:

1. Contraindication to any drug contained in the chemotherapy regimen or to any of their excipients
2. T-cell lymphoma
3. Diagnosis of any second malignancy within the last 5 years
4. Prior history of organ transplantation or other cause of severe immunodeficiency
5. History of heart disease and/or impaired cardiac function (ECG QTc>450msec, congenital long QT syndrome, history of ventricular tachyarrhythmia, ventricular fibrillation, congestive heart failure NYHA III/IV, uncontrolled hypertension).
6. Known HIV or HTLV-1 infection, positive serology to HB surface antigen [HBsAg] or total HB core antibody [anti-HB-c]) and Hepatitis C (Hepatitis C virus [HCV] antibody) not older than 4 weeks
7. Inclusion in another experimental anti-cancer drug therapy*
8. Impossibility to follow the calendar of exams because of geographic, social or psychological reasons
9. Patient under measure of legal protection
10. No social security *For ethical reasons, the exclusion period within which the patient cannot be included in another trial will not be defined but discussed on a case to case basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-09-18 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of lenalidomide in combination with rituximab in relapsed/refractory PCNSL as measured by the objective response rate (CR + uCR + PR) at the end of the 8 cycles of induction therapy. | 33 months
  The objective response rate (CR+uCR+PR) will be evaluated according to the IPCG (International Primary CNS lymphoma Collaborative Group) recommendations. Patients will have an cerebral MRI, an ophthalmological examination and a lumbar puncture at several times.

SECONDARY OUTCOMES:
The safety of the association during induction and maintenance therapy in a population of PCNSL (NCI V4) | 56 months
The duration of response | 56 months
Progressive Free Survival at one year from the date of inclusion to the date of progression of the disease or death | 56 months
Overall Survival from the date of inclusion to the date of death | 56 months
Quality of life using QLQ-C30 EORTC (European Organization for Research and Treatment of Cancer) questionnaire | 20 months

OTHER OUTCOMES:
Exploration of T cells and NK (Natural Killer) cells populations in PCNSL before and after treatment to correlate possible changes of these populations with therapeutic response | 33 months
  Pilot exploration of T cells and NK cells populations in PCNSL before and after treatment with the combination of lenalidomide-rituximab and to correlate possible changes of these populations with therapeutic response

CONTACTS AND LOCATIONS:
Overall Officials: Carole SOUSSAIN, MD, Principal Investigator — Institut Curie - Hopital Rene Huguenin
Locations (12):
- France (12):
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - CHU Estaing, Clermont-Ferrand, Auvergne
  - CHU Bretonneau - Centre Henry Kaplan, Tours, Centre-Val de Loire
  - Institut Bergonié, Bordeaux, Gironde
  - Chu Michallon, Grenoble, Isère
  - Hôpital Central, Nancy, Lorraine
  - CHRU Lille - Hôpital Claude Huriez, Lille, Nord
  - Centre Henri Becquerel, Rouen, Seine Maritime
  - CHU Amiens -Hôpital Sud, Amiens, Somme
  - Chu La Timone, Marseille
  - Hôpital de la Pitié Salpétrière, Paris, Île-de-France Region
  - Institut curie - Hôpital René Huguenin, Saint-Cloud, Île-de-France Region

REFERENCES:
- [Result] Ghesquieres H, Chevrier M, Laadhari M, Chinot O, Choquet S, Molucon-Chabrot C, Beauchesne P, Gressin R, Morschhauser F, Schmitt A, Gyan E, Hoang-Xuan K, Nicolas-Virelizier E, Cassoux N, Touitou V, Le Garff-Tavernier M, Savignoni A, Turbiez I, Soumelis V, Houillier C, Soussain C. Lenalidomide in combination with intravenous rituximab (REVRI) in relapsed/refractory primary CNS lymphoma or primary intraocular lymphoma: a multicenter prospective 'proof of concept' phase II study of the French Oculo-Cerebral lymphoma (LOC) Network and the Lymphoma Study Association (LYSA)dagger. Ann Oncol. 2019 Apr 1;30(4):621-628. doi: 10.1093/annonc/mdz032. PMID 30698644
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30698644/